CLINICAL TRIAL: NCT02435784
Title: The Two-Way Communication Checklist (2-COM) in First Episode Psychosis Patients in Hong Kong: an Open Label Randomized Controlled Trial
Brief Title: The Two-Way Communication Checklist (2-COM) in First Episode Psychosis Patients in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chau Wing Leong, RN(Psy), Kwai Chung Hospital, Hong Kong, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UW 15-170
Record Dates: First submitted 2015-04-22; First posted 2015-05-06 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia; Communication
Keywords: 2-COM
MeSH Terms: conditions — Schizophrenia; Communication | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2-COM group (Active Comparator): Patients will use the Two-Way Communication Checklist (2-COM) once in a psychiatric consultation.
  Interventions: Other: The Two-Way Communication Checklist
- TAU group (Placebo Comparator): Treatment as usual (TAU) group.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: The Two-Way Communication Checklist — The Two-Way Communication Checklist (2-COM) is a communication tool developed by Van Os et al. (2002). It aims to provide an opportunity for patients to voice their needs and problem to minimize the discrepancy and miscommunication between patient and professional carer. 2-COM questionnaire was designed to give patients while they are waiting for consultation. Patients can either tick yes or no in the questionnaire to decide which the perceived problems are and which needs they want to discuss with the clinician. During the consultation, the ticked items would be discussed.
  Other Names: 2-COM
  Arms: 2-COM group
Other: Treatment as usual — Patients will attend a psychiatric consultation as usual.
  Other Names: TAU
  Arms: TAU group

SUMMARY:
The Two-Way Communication Checklist (2-COM) is a communication tool developed by van Os et al. (2002). It aims to provide an opportunity for patients to voice their needs and problem to minimize the discrepancy and miscommunication between patient and professional carer. In this randomized controlled trial, the investigators aim to examine whether using 2-COM checklist would lead to improvement in first episode psychosis patient's overall satisfaction, change in treatment option in clinicians and consultation time.

DETAILED DESCRIPTION:
Communication is at the heart of psychiatric practice. Good communication has positive impact on treatment, treatment satisfaction and treatment adherence. However, different characteristics of psychosis barricade the communication between clinicians and patients. Consequently, the divergent views of needs of care between patients and clinicians may be established due to miscommunication. Such divergence may barricade the planning and the outcome of treatment.

In Hong Kong, the core psychiatric services as well as early intervention for first episode psychosis patients are provided by psychiatric outpatient clinics. Mental health services in Hong Kong are overwhelmed by large demands of the services and inadequate mental health care workforce such as low psychiatrists-to-population ratio and psychiatric nurse-to-population ratio. The large demands of services and inadequate mental health care workforce restrained the services' quality. In some busy psychiatric outpatient clinic, a clinician needs to consult 30 patients in a 3-hour session. Hui et al. (2008) study showed that the mean consultation time in one of the general psychiatric outpatient clinic in Hong Kong is 5.8 minutes.

To sum up, a cost-effectiveness instrument is in need for the early intervention psychiatric outpatient clinic in Hong Kong. The instrument has to reduce the needs' divergence, communication between clinicians and patients, and enhance the patients' involvement of clinical decision-making in the rushed psychiatric consultation. The Two-Way Communication Checklist (2-COM) may satisfy the demand.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they meet the following criteria:

1. attended the EASY service;
2. were diagnosed with schizophrenia ,schizoaffective disorder or schizophreniform disorder according to ICD-10;
3. were age between 15-64;
4. were able to complete the informed consent.

Exclusion Criteria:

Patients will be excluded if they meet the following criteria:

1. had history of substance misuse;
2. had history of intellectual disability;
3. were non- Chinese speaking patients
4. had violent risk
5. had suicidal risk

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Satisfaction level (patient satisfaction questionnaire) | within 30 minutes after a psychiatric consultation
  A patient satisfaction questionnaire as used in Hui et al. (2008) was adopted in this study. This was a self-administered questionnaire rated on a 5-point Likert scale (1 = very satisfactory to 5 = very unsatisfactory). The questionnaire consisted of 2 parts. Part A has 6 items concerning the perceived attitude of the clinician (subscale score range, 6-30). Part B has 11 items concerning communication with the clinician (subscale score range, 11-55). The higher score indicates the higher satisfaction.

SECONDARY OUTCOMES:
Change of treatment (checklist) | within 30 minutes after a psychiatric consultation
  A checklist that measured change in treatment was adopted. This checklist included 4 items which will be rated on a dichotomous selection (yes/no) by clinician. The 4 items are related to the change of medication, providing information about treatment, involvement of other members of the care team and professional support services.
Consultation time | From the time of patients' entering the consultation room till leaving the consultation room in a psychiatric consultation, up to 5 hours
  The consultation time will be counted between patients' entering and leaving the consultation room by a stopwatch.

CONTACTS AND LOCATIONS:
Overall Officials: Wing Leong Chau, RN(Psy), Principal Investigator — Kwai Chung Hospital
Locations (1):
- EASY Clinic, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Lam MM, Pearson V, Ng RM, Chiu CP, Law CW, Chen EY. What does recovery from psychosis mean? Perceptions of young first-episode patients. Int J Soc Psychiatry. 2011 Nov;57(6):580-7. doi: 10.1177/0020764010374418. Epub 2010 Jul 5. PMID 20603266
- [Background] Hui, C. L. M., Wong, G. H. Y., Lam, C. Y. K., Chow, P. P. L. & Chen, E. Y. H. (2008). Patients-clinician communication and needs identification for outpatients with schizophrenia in Hong Kong: role of the 2-COM instrument. Hong Kong Journal of Psychiatry, 18(2), 69-74.
- [Background] Chan KK, Mak WW. The mediating role of self-stigma and unmet needs on the recovery of people with schizophrenia living in the community. Qual Life Res. 2014 Nov;23(9):2559-68. doi: 10.1007/s11136-014-0695-7. Epub 2014 Apr 23. PMID 24756436
- [Background] Wong GH, Hui CL, Wong DY, Tang JY, Chang WC, Chan SK, Lee EH, Xu JQ, Lin JJ, Lai DC, Tam W, Kok J, Chung DW, Hung SF, Chen EY. Developments in early intervention for psychosis in Hong Kong. East Asian Arch Psychiatry. 2012 Sep;22(3):100-4. PMID 23019282
- See also: Previous 2-COM studies — http://2coms.homestead.com/